CLINICAL TRIAL: NCT03243591
Title: Impact of Oral Hygiene Gels on Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0388-17-EP
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Mucositis
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, double-blind, single center
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Gels are in coded opaque tubes created at the manufacturer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Livionex gel (Active Comparator): Brushing area of mucositis with Livionex gel for 30 days
  Interventions: Other: Livionex gel
- Aquafresh gel (Active Comparator): Brushing area of mucositis with Aquafresh gel for 30 days
  Interventions: Other: Aquafresh gel

INTERVENTIONS:
Other: Livionex gel — Brushing area of mucositis with gel
  Other Names: Aquafresh gel
  Arms: Livionex gel
Other: Aquafresh gel — Aquafresh gel
  Arms: Aquafresh gel

SUMMARY:
Peri-implant mucositis is abnormal inflammation occurring around dental implants, increasing the risk of loss of bone support. The purpose of this study is to evaluate the impact of brushing the bacterial biofilm at the implant-mucosa interface with one of two, commercially-available dental gels over a 30-day period on amounts of biofilm and indices of mucosal inflammation. Adult subjects (> 19 years old) will be invited to consent if they have at least one dental implant displaying mucositis defined as Gingivitis Index of 2 or greater, no dental treatment in the previous 30 days, capable of normal toothbrushing, and no Sjogrens disease, immunodeficiency, pregnancy, poorly-controlled diabetes, or regular systemic antibiotics, anti-inflammatory drugs or immune suppressants. Ten patients in each tooth gel group will be instructed to apply a pea size amount of dentifrice brushing the implant and mucosa 2 times daily for 30 days. Baseline and 30-day examinations will be conducted to record Gingivitis Index, Plaque Index, probing depths, clinical photo, crevicular fluid, and adverse events.

DETAILED DESCRIPTION:
This will be a prospective, randomized, controlled, double-blind, single center study. Once eligibility has been determined, up to 21 Subjects will be enrolled. Subjects will be randomly assigned in a 1:1 ratio to treat with either Livionex Dental Gel (a plaque control gel that is safe for ingestion and is currently sold by Livionex Inc.) or the control Aquafresh toothpaste. Each study visit will last 30 minutes.

The soft tissue around the dental implant will be observed at baseline and after 30 days for inflammation using the Gingivitis Index and probed with a UNC 15 periodontol probe for pocket depth and bleeding. A photograph will be taken of the most inflamed side of the implant. Plaque will be stained with oral hygiene staining rinse and evaluated for Plaque Index. Finally, a paper strip will be inserted between the gingiva and implant on facial and lingual sides for 30 seconds each.

GINGIVITIS INDEX: Gingivitis score (GI)= Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation slight change in color and little change in texture 2 = Moderate inflammation moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding. GI scored=sum of GI scores divided by the number of sites (gingival gum line around the tooth) scored.

PLAQUE INDEX Using Quigley Staining Hein Method with Turesky Modification:Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth. Plaque score = sum of all scores divided by the number of sites (teeth) scored.

Each patients will be instructed to brush around the implant with a pea size amount of dentifrice provided, twice daily for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* history of 5 mm+ pocket bleeding on probing around implant

Exclusion Criteria:

* dental treatment of implant in previous 30 days
* Sjogrens disease
* immunodeficiencies (e.g. AIDS)
* poorly-controlled diabetes
* regular use of antibiotics, anti-inflammatory drugs or immune suppressants

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Gingival Index | 30 days
  Level of clinical inflammation around dental implant

SECONDARY OUTCOMES:
Plaque Index | 30 days
  Amount of biofilm around dental implant
Crevicular Fluid Biomarkers | 30 days
  Fluid from around implant measured for inflammation markers with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Reinhardt, DDS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No